CLINICAL TRIAL: NCT01128517
Title: Does Maternal Education on Complementary Feeding Have an Impact on Infant Nutritional Status in Low Middle-income Households? A Community Based Randomized Interventional Study in Karachi, Pakistan.
Brief Title: Maternal Education on Complementary Feeding and Infant Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Ali Faisal Saleem, The Aga Khan University Hospital, Karachi. Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MECF
Record Dates: First submitted 2010-05-17; First posted 2010-05-24 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2010-04

CONDITIONS: Growth
Keywords: Maternal education; Complementary food; Infant growth
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bahavioral (Experimental): Education about complementary food given to mothers
  Interventions: Behavioral: Maternal education on complementary feeding; Behavioral: Education

INTERVENTIONS:
Behavioral: Maternal education on complementary feeding — CF education to the mothers in intervention arm.
  * Ten important key messages developed based on recommended practices (WHO/UNICEF, 2000 & 2006).
  * First session --> cover the importance of breast feeding, its continuation for whole two years, hand washing, hygiene and importance of CF initiation at 6 months of age.
  * Second session -->breastfeeding promotion, complementary food consistency, initial complementary food selection and age related complementary food education.
  * Third session --> previous sessions recall. protein based and iron rich food encouragement.
  * The control arm continue to be benefited from the lady health workers program, while breastfeeding promotion would be provided to control arm
  Other Names: Packaged teaching education to mothers on different visits
Behavioral: Education — Maternal education on complementary food
  Other Names: Education to mothers given in three teaching modules.

SUMMARY:
Overall Objective

• To evaluate impact of maternal educational strategies (teaching sessions by trained lady health workers, verbal, pictorial and demonstrative) regarding appropriate complementary foods of infants, and assess their impact on nutritional status of after six months of educational intervention.

Specific objective • To determine the impact of maternal educational strategies regarding complementary foods by assessing baseline weight, height and mid - upper arm circumference at 2.5 - 5 month of age and then comparing it at 3, 6 and 9 months after enrollment.

(Hypothesis; the investigators hypothesize that there will be a gain of 250 gram weight, 0.5 cm in length and 0.5 cm in MUAC in infants whose mothers received the special education module for complementary feeding, as compare to the children whose mothers doesn't receive education on complementary food.

Secondary objective

• To determine the impact of maternal educational strategies regarding complementary foods by assessing morbidity (number of diarrhea and ARI episodes, at 2.5 - 5 month of age and at then reporting at 3, 6 and 9 months after enrollment).

(Hypothesis; the investigators hypothesize that there will be 10% decrease in incidence of diarrhea episodes and ARI episodes in infants whose mother received the special education module for complementary feeding, as compare to the children whose mothers doesn't receive education on complementary food).

ARI can be define as per IMCI guidelines. Increase breathing rate (age specific) along with cough, cold and or wheezing.

DETAILED DESCRIPTION:
Study population The study will be conducting in Bhainse colony (BC), Karachi. This is a periurban community area, and catering population mainly belonging to low - middle income households. The study population would be the mothers (having infant of 2.5 - 5 months of age) and their infants in these two study areas.

Inclusion Criteria;

* Infants aged 2.5 - 5 months; who are either exclusively breast feed or partially breast feed but have not started complementary feeding or have recently started complementary food (less than 1 week)
* Informed consent Exclusion Criteria;
* Infants found below 5th percentile on weight for age CDC growth charts 23 at baseline will be excluded.
* History of two or more hospital admissions for more than 7 days each
* Presence of serious congenital anomalies (cleft palate, congenital heart disease, neural tube defect) or other chronic conditions impairing feeding (e.g. cerebral palsy)
* Presence of acute illness requiring urgent hospitalization
* Infants from families of very low socioeconomic status where adequate calorie-provision is constrained (assessed by a questionnaire on household possessions of items such as mobile phone, bicycle or other vehicle, TV, cemented construction, fuel used for cooking - wood or gas/LPG)
* Infant already enrolled in any trial with a nutritional intervention will be excluded.
* Infants who at initial clinical examination are found to be severely anemic.

Data outcome measures Measuring Weight, height and Mid-upper arm circumference The investigators measure serial height, weight and mid-upper arm circumference (MUAC) for each subject at enrollment and subsequently in each visit. Each infant will be measured four times during the study enrollment.

* Height will be measured twice and the results averaged. Duplicate measures that exceed predefined allowable variation will be resolved by the field supervisor, e.g., by returning to the site with the interviewer to repeat the measurements. The height of infants will be measured (to the nearest 0.1 cm) in the recumbent position using a board with a fixed head and sliding foot piece.
* Weight will be measured to the nearest 0.1 kg using a scale that is calibrated daily.
* MUAC will be measure twice each time by using measuring tape. All anthropometric measurements will be taken three times (in each visit) and the mean of the measurements will counted as valid value. Each of the anthropometric indices will be expressed in standard deviation units (SD) from the median of the NCHS/CDC/WHO International Reference Population. Methods are adapted from How to Weigh and Measure Children: Assessing the Nutritional Status of Young Children in Household Surveys, United Nations Department of Technical Cooperation for Development and Statistical Office, 1986. The height and weight measurements will later converted into WAZ, WHZ and HAZ score and the difference in both groups will be analyzed.

  * ARI will be measured through standard IMCI guidelines. ARI could be assess by the physician's visit and treatment prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 2.5 - 5 months; who are either exclusively breast feed or partially breast feed but have not started complementary feeding or have recently started complementary food (less than 1 week)
* Informed consent

Exclusion Criteria:

* Infants found below 5th percentile on weight for age CDC growth charts at baseline will be excluded
* History of two or more hospital admissions for more than 7 days each
* Presence of serious congenital anomalies (cleft palate, congenital heart disease, neural tube defect) or other chronic conditions impairing feeding (e.g. cerebral palsy)
* Presence of acute illness requiring urgent hospitalization
* Infants from families of very low socioeconomic status where adequate calorie-provision is constrained (assessed by a questionnaire on household possessions of items such as mobile phone, bicycle or other vehicle, TV, cemented construction, fuel used for cooking - wood or gas/LPG)
* Infant already enrolled in any trial with a nutritional intervention will be excluded
* Infants who at initial clinical examination are found to be severely anemic

Ages: 3 Months to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Nutritional status | 7.5 month
  Height, Weight and Mid Upper Arm circumference

SECONDARY OUTCOMES:
Diarrhea episodes | 7.5 months
  Diarrhea episodes during the study period.
Z score (HAZ, WAZ and WHZ scores) | 7.5 months
  Z scores (wasting, stunting will be measured and compared in between interventional and control group.
ARI | 7.5 months
  ARI will be asses by using standard IMCI guidelines, and/or physician prescription and medications prescribed to the infant.

CONTACTS AND LOCATIONS:
Overall Officials: Ali F Saleem, MBBS, Principal Investigator — The Aga Khan University Hospital, Karachi, Pakistan
Locations (1):
- Bhainse colony, Karachi, Sindh, Pakistan